CLINICAL TRIAL: NCT04060446
Title: Effects of Filter Ventilation on Sensory Response, Smoking Topography, and Inhalation (COMET 2 2.1)
Brief Title: Effects of Filter Ventilation on Sensory Response, Smoking Topography, and Inhalation in Current Every Day Cigarette Smokers
Status: Completed | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: I 68718; NCI-2019-04530 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 68718 (Other: Roswell Park Cancer Institute); P01CA217806 (NIH); P30CA016056 (NIH)
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Cigarette Smoker; Current Every Day Smoker
MeSH Terms: interventions — Equipment and Supplies; Smoking Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (smoke cigarettes): Patients smoke 5 cigarettes separated by 30 minute washout periods. Between 48 hours and 1 week later, patients smoke another 5 cigarettes separated by 30 minute washout period with CReSSMicro topography measurement device and BioRadio device for recording inhalation patterns.
  Interventions: Device: Medical Device; Other: Questionnaire Administration; Behavioral: Tobacco Smoking

INTERVENTIONS:
Device: Medical Device — Smoke cigarettes with CReSSMicro topography measurement device and BioRadio device
  Other Names: Device; Medical Devices
Other: Questionnaire Administration — Ancillary studies
Behavioral: Tobacco Smoking — Smoke cigarettes
  Other Names: Smoking

SUMMARY:
This trial examines the effects of filter ventilation on sensory response, smoking topography, and inhalation in current every day cigarette smokers. The physical design features of cigarettes directly impact their appeal by influencing cognitive and sensory perceptions. The introduction of a now common design feature, filter ventilation, has led to greater public harm than benefit because of the potential for greater toxicity while enhancing product appeal among smokers. Ventilated cigarettes dilute smoke, which promotes perceptions of ?smoothness? and therefore lower health risk, contributing to the overall appeal of these products. The purpose of this study is to assess whether removing ventilation from cigarette filters lowers cigarette product appeal among smokers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the link between marketing proxies for filter ventilation (product descriptors, packaging) and risk beliefs.

OUTLINE:

Patients smoke 5 cigarettes separated by 30 minute washout periods. Between 48 hours and 1 week later, patients smoke another 5 cigarettes separated by 30 minute washout period with CReSSMicro topography measurement device and BioRadio device for recording inhalation patterns.

ELIGIBILITY:
Inclusion Criteria:

* Currently smoking daily at least 5 cigarettes per day for at least one year
* Primarily using factory-made filtered cigarettes with filter ventilation
* Fair and above physical health
* Fair and above mental health
* Not actively trying to quit smoking or planning to quit in the next 30 days
* Able to converse, read, and write in English
* No alcohol or illegal drug use
* Not pregnant or breastfeeding

Exclusion Criteria:

* Currently smoking daily less than 5 cigarettes per day for at least one year
* Using roll-your-own cigarettes or unventilated filter cigarettes
* Currently using any other tobacco product daily
* Actively trying to quit smoking or planning to quit in the next 30 days
* Not able to converse, read, and write in English
* Adults unable to consent
* Prisoners
* Poor physical health by self report
* Poor mental health by self report
* Alcohol and illegal drug use
* Pregnant or breastfeeding by self report

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients currently smoking daily at least 5 cigarettes per day for at least one year
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Modified Cigarette Evaluation Questionnaire | Up to 210 minutes
  Scored using an established algorithm. This results in 3 subscales (psychological reward, relief, reward) and 2 single items (aversion, respiratory sensation).

SECONDARY OUTCOMES:
Carbon monoxide (CO) boost | Up to 210 minutes
  Defined as the difference between pre-smoking exhaled CO and postsmoking exhaled CO.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J O'Connor, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States